CLINICAL TRIAL: NCT06631846
Title: Efficacy of Music Therapy and Mindfulness Meditation on Hemodynamic Variables and Mental Health Among Coronary Artery Bypass Graft Patients
Brief Title: Music Therapy and Mindfulness Meditation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Imtiyaz Ali Mir, Principal Investigator, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Music Therapy and Mindfulness
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Bypass Graft Surgery Patients
Keywords: Coronary Artery Bypass Graft Patients; Hemodynamic Variables; Mental Health; Music Therapy; Mindfulness Meditation; Anxiety; Depression; Quality of life
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders; Depression | interventions — Music Therapy; Mindfulness; Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Music therapy (Experimental)
  Interventions: Other: Music therapy
- Mindfulness meditation (Experimental)
  Interventions: Other: Mindfulness meditation
- Combination of music therapy and mindfulness meditation (Experimental)
  Interventions: Other: Music therapy and mindfulness meditation
- Conventional phase-1 cardaic rehabilitation (Active Comparator)
  Interventions: Other: Cardiac rehabilitation

INTERVENTIONS:
Other: Music therapy — Participants in the music therapy group (MTG) will be comfortably lying on the bed in a reclined position of 30-45 degrees. Using a headphone, participants will be instructed to select a volume that is comfortable to their ears and listen to the music titled as "The Best Relaxing Piano and Flute Music Ever" which will be played for 30-minutes every day for 1-week. Patients will be encouraged to focus on the music and let it fill their senses.
  Arms: Music therapy
Other: Mindfulness meditation — Mindfulness meditation group (MGT)will be listening to audio of Guided Mindfulness Meditation Series 1 by Jon Kabat-Zinn. Similar to MTG, participants in MMG will be lying on the bed in a reclined position of 30-45 degrees. A headphone to listen to the audio of guided MM will be provided to all the participants. Participants will begin with relaxation technique by focusing on deep breathing to help calm their body and mind. This will be followed by focusing on the present moment, letting go of any thoughts or distractions that come up. Participants can focus on their breath, bodily sensations, or a specific object in their environment. Finally, the session will end by expressing a gratitude for their body and mind and setting an intention to carry the feelings of relaxation and mindfulness with them throughout the day. Similar to MTG, MMG will engage in 30-minutes of MM every day for 1-week.
  Arms: Mindfulness meditation
Other: Music therapy and mindfulness meditation — Music therapy and mindfulness meditation group will be receiving both music therapy and mindfulness meditation in the same body position as MTG and MMG. Firstly, participants will listen to MT for 30-minutes followed by MM for another 30-minutes. In between the 2 interventions, a 15-minute of break will be provided to all participants. Intervention will be carried out every day for 1-week.
  Arms: Combination of music therapy and mindfulness meditation
Other: Cardiac rehabilitation — Control Group will not receive any other therapy except the conventional post-operative cardiac rehabilitation. Other 3 intervention groups will also be participating in the usual cardiac rehabilitation program. Cardiac rehabilitation will be conducted during phase I, where rehabilitation will focus on early mobilization and ambulation of participants with a target heart rate of resting heart rate + 30 beats, with the non-strenuous exercises in the bed or at the bedside, focusing on a range of motion and limiting hospital deconditioning.
  Arms: Conventional phase-1 cardaic rehabilitation

SUMMARY:
Coronary artery bypass graft surgery (CABG) involves bypassing a blocked artery with a healthy blood vessel elsewhere from body allowing the blood flow to be restored to heart. Most patients after CABG surgery have hemodynamic instability such as elevated blood pressure (BP) and low heart rate variability (HRV). High BP could be due pain, stress, and withdrawal of BP medications, which patient used to take preoperatively. BP progressively increases within 24 hours, postoperatively, and daytime systolic and diastolic BP may remain elevated for =14 weeks after CABG, while lower HRV may take 6 months to recover after CABG. In addition, these patients suffer from anxiety and depression which is associated with poor mental health that can create significant challenges and barriers for patients in making and sustaining important behavioral and lifestyle modifications. Non-pharmacological interventions such as music therapy (MT) and mindfulness meditation (MM) have been successfully used to manage anxiety and depression among patients undergone various surgeries, but there is scarcity in the current literature with regards to investigating the combined effect of MT and MM on anxiety and depression in CABG patients. Furthermore, the cumulative effect of these 2 interventions on hemodynamic variables is not well established. Therefore, this study aims to bridge these gaps and develop an interventional protocol that can improve the hemodynamic stability and mental health of CABG patients.

DETAILED DESCRIPTION:
Coronary artery bypass graft surgery (CABG) is an invasive procedure to treat coronary artery disease (CAD). The blocked section of the coronary artery is bypassed by using a healthy blood vessel or graft elsewhere from our body allowing the blood flow to be restored to heart. After CABG surgery, these patients encounter the problems of hemodynamic instability such as high blood pressure (BP) and low heart rate variability (HRV).

There are multiple reasons why BP increases, including pain, stress, and withdrawal of BP medications, which patient was receiving preoperatively. Typically, the BP progressively increases within 24 hours, postoperatively, and daytime systolic and diastolic BP may remain elevated for 14 weeks after CABG. In addition, nocturnal BP dipping returns to normal progressively but incompletely 14 weeks after CABG. HRV is found to lower after the CABG surgery, and it might take 6 months for the HRV to recover. The percentage of HRV after 7 days of CABG surgery was found to be 51.8%, 19.6% after 3 months, and 12.7% after 6 months.

Patients in the post-operative phase also suffer from anxiety and depression due to fear of death, pain, confusion, and sleeping disorders that can lead to poor functional mobility and quality of life. If anxiety and depression is not addressed in these patients, it could lead to major adverse cardiovascular and cerebrovascular events like myocardial infarction and stroke.

Anxiety, depression, and stress have been shown to increase the production of inflammatory cytokines such as interleukin-6 (IL-6), and elevation of C-reactive protein (CRP). Both IL-6 and CRP can affect vascular tone by promoting the production of endothelin-1 and impairing the production of nitric oxide, a potent vasodilator which will lead to hemodynamic instability by causing vasoconstriction and reduced cardiac output. The cytokines can activate the coagulation system by increasing the expression of tissue factor and reducing the production of anticoagulant factors such as thrombomodulin. Furthermore, stress can also lead to increased sympathetic nervous system activity, which can further exacerbate the effects of IL-6 and CRP on hemodynamic instability. Sympathetic activation can cause vasoconstriction and increase heart rate and contractility, leading to increased myocardial oxygen demand and reduced coronary perfusion.

The hypothalamic-pituitary-adrenal (HPA) axis and the sympathetic-adrenomedullary pathways (SAP) which activate the sympathetic nervous system, are major stress response systems in the body that regulate the release of cortisol, and stress hormones. These hormones can impair fibrinolysis by reducing the production of plasminogen activators and increasing the production of plasminogen activator inhibitors, leading to an increase in heart rate, blood pressure, and cardiac output. These changes can contribute to hemodynamic instability after CABG surgery. A study found that patients with post-traumatic stress disorder had higher levels of cortisol and plasminogen activator inhibitor-1 compared to controls, suggesting a link between stress, and altered fibrinolysis. A reviews based on various epidemiological studies and clinical trials investigated the association between stress and thrombosis and study concluded that acute and chronic stress can increase the risk of thrombosis, including activation of the sympathetic nervous system, increased platelet activation, and alterations in blood coagulation and fibrinolysis, which may further lead to an increased risk of hemodynamic instability after CABG surgery. Dysregulation of the HPA axis and SAP have been implicated in the development and progression of coronary artery disease (CAD). In addition, dysregulation of both these systems can contribute to a state of chronic stress in depressed individuals, which can have negative effects on physical and mental health and increase the risk of developing cardiovascular disease, as well as worsen the symptoms of depression and anxiety.

A study showed that 30% to 40% of post CABG surgery patients experience psychological disorder like depression and anxiety which increase the rate of morbidity even after years of discharge. A meta-analysis found that nearly one-third of CABG patients were depressed before surgery and their symptoms significantly improved after the surgery. However, the study also indicated that approximately one-fifth of those who undergo CABG remain depressed or develop new depression. A 2-year prospective follow-up study found that post-CABG patients suffered from chronic depression and had a significantly higher incidence of cardiac events and hospitalization rates compared to patients without depressive symptoms. Therefore, it is important to address these issues in patients after CABG surgery, which would potentially influence the outcomes of the hemodynamic variables. Non-pharmacological intervention like music therapy (MT), and mindfulness meditation (MM) have been successfully used to manage anxiety and depression among patients with different surgeries in post-operative phase.

There have been many studies conducted to explore the potential benefits of MT in reducing stress and anxiety during surgery and decreasing the need for anaesthesia focused on patients undergoing elective orthopaedic surgery and effect of MT on open-hernia surgery. Both these studies aimed to assess the stress levels and anaesthetic drug requirements of patients before and after MT intervention. Authors provided valuable insights for developing effective intervention that can assist patients in managing stress and anxiety associated with surgery, and potentially decrease their reliance on anaesthesia. Furthermore, compared to the control group, individuals who listened to music for 30-minutes shows increased levels of oxytocin.

A recent systematic review found that music not only affects the patients' emotional and psychological well-being via the autonomic nervous system (ANS), but it can also have a potential impact on cardiovascular variables, including HRV, heart rate (HR), respiration rate (RR), and BP. Research has established that HRV is a biomarker that reflects the activity of the ANS. Therefore, MT can be a promising intervention tool to regulate both HRV and ANS.

MM originated from Buddhism and has been practiced for over 2550 years. In early 1960s, it was introduced to the Western psychology and healthcare sectors. This non-pharmacological intervention has since evolved and been extensively reviewed, with findings indicating that it has a significantly positive impact on psychological health. Specifically, it has been found to reduce symptoms of anxiety, depression, rumination, psychological distress, cognitive disorganization, post-traumatic avoidance symptoms, and medical symptoms. It also increases the positive sense of spirituality, empathy, sense of cohesion, and self-compassion, and improve quality of life, satisfaction of life in clinical and non-clinically patients with psychosocial and existential distress.

According to Kabat-Zinn, mindfulness-based stress reduction could significantly reduce BP in patients with coronary heart disease by an average of 8 mmHg after only 8-weeks of treatment. Similarly, a study found that 4-weeks of mindfulness-based cognitive therapy resulted in improved symptoms for patients with chronic heart failure. The effects of an 8-week MM program on inflammatory markers were examined in healthy adults. The study found that the MM group had lower levels of the inflammatory marker IL-6 compared to a control group. This highlights the potential benefits of mindfulness-based intervention for improving health outcomes by reducing inflammatory markers.

Another study investigated the effect of MM on immunological function in women diagnosed with breast cancer. Researchers discovered significant improvements in women's immune function, with lower levels of pro inflammatory cytokines and decreased production of IL-6, compared to the active control group. Additionally, notable enhancements in patients' psychological well-being, including reduced levels of anxiety, depression, and stress was noticed.

A recent meta-analysis on MM reported significantly decrease cortisol levels in patients at risk of various health problems, such as cardiovascular disease, depression, and anxiety. Furthermore, the use of MM intervention was found to have a beneficial impact on the HRV, which is a primary time domain measure for vagal tone.

In conclusion, both MT and MM have been found to induce changes in the prefrontal cortex region of the brain. Specifically, these changes are observed in the limbic pathway, which is highly responsive to human behaviour and emotional changes, and plays an important role in the regulation of ANS. Additionally, both interventions positively influence the cardiac autonomic system and hemodynamic variables through the stimulation of the vagus nerve, which has been shown to have direct advantages in managing cardiovascular health by reducing anxiety and depression.

At present, exercise-based cardiac rehabilitation is the single recommended secondary prevention strategy for cardiac patients that aims to address anxiety and psychosocial wellbeing, and there is a critical gap to address psychosocial needs of cardiac patients, particularly in CABG patients. Poor mental health and associated negative emotions can create significant challenges and barriers for patients in making and sustaining important behavioral and lifestyle modifications. Although MT and MM individually are reported to be effective in managing the psychological problems such as anxiety and depression, but there is scarcity in the current literature with regards to investigating the cumulative and combined effect of these 2 interventions. Therefore, this study aims to bridge this gap and develop an interventional protocol that can address and improve the mental health and overall quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Both gender of age 18 and above
* Undergone isolated CABG
* Ejection fraction ≥ 50%
* Hemodynamically stable
* Willing to participate in this study

Exclusion Criteria:

* Participants with atrial fibrillation
* Hearing abnormalities
* Cardiovascular diseases other than coronary artery disease, respiratory diseases, and any neurological/musculoskeletal problems that will restrict eligible participants to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure will be measured using a calibrated digital BP measuring monitor among 48 participants after CABG. | At baseline before beggining intervention and post-intervention at the end of1-week.
Diastolic blood pressure will be measured using a calibrated digital BP measuring monitor among 48 participants after CABG. | At baseline before beggining intervention and post-intervention at the end of 1-week.
Heart rate variability will be measured using a standard portable 12 lead ECG machine among 48 participants after CABG. | At baseline before beggining intervention and post-intervention at the end of 1-week.
Anxiety will be measured utilizing Beck Anxiety Inventory (BAI), which consists of 21 self-reported items to assess the intensity of physical and cognitive anxiety symptoms during the past week among 48 participants after CABG. | At baseline before beggining intervention and post-intervention at the end of 1-week.
Depression will be measured utilizing Beck Depression Inventory (BDI), which consists of 21 self-reported items to assess the characteristic attitudes and symptoms of depression during the past week among 48 participants after CABG. | At baseline before beggining intervention and post-intervention at the end of 1-week.

SECONDARY OUTCOMES:
Quality of life will be measured using Short Form 12 Health Survey (SF-12), which consisted of 12 short from items measuring the extent to which physical or emotional problems interfere with social activities among 48 participants after CABG. | At baseline before beggining intervention and post-intervention at the end of 1-week.

IPD SHARING:
Plan to Share IPD: No